CLINICAL TRIAL: NCT00049751
Title: A Multicenter Study of the Safety of Human Anti-TNF Monoclonal Antibody D2E7 in Subjects With Active Rheumatoid Arthritis
Brief Title: Study of Human Anti-TNF Monoclonal Antibody D2E7 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-498
Record Dates: First submitted 2002-11-13; First posted 2002-11-14 (Estimated); Last update posted 2006-08-15 (Estimated); Status verified 2006-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

INTERVENTIONS:
Drug: Adalimumab

SUMMARY:
The purpose of the study is to evaluate safety by collecting serious adverse events in subjects with moderately to severely active rheumatoid arthritis who are unable to obtain etanercept and who have failed one or more prior disease-modifying antirheumatic drugs (DMARDs).

ELIGIBILITY:
Inclusion:

* Subjects must meet ACR criteria for diagnosis of RA for at least 3 months, must meet ACR Functional Class I, II or III (1992 criteria) and must have a confirmed diagnosis of active moderate to severe rheumatoid arthritis as defined by 6 or more swollen joints and 9 or more tender joints;
* must also have DAS of 3.2 or greater at study entry,
* normal laboratory parameters and ESR >20,
* satisfactory response or intolerance to one or more prior DMARDs and
* be willing and able to give informed consent.

Exclusion:

* Previous treatment with total lymphoid irradiation or anti-CD4 or CAMPATH 1H monoclonal antibodies resulting in persistent CD4 lymphopenia,
* history of acute inflammatory joint disease other than RA,
* prior treatment with cyclophosphamide or chlorambucil,
* prior treatment with intravenous immunoglobulin within 70 days,
* history of malignant lymphoma,
* history of uncontrolled diabetes,
* unstable ischemic heart disease,
* active inflammatory bowel disease,
* active peptic ulcer disease or stroke,
* positive HIV status,
* positive serology for Hepatitis B or C,
* no previous history of tuberculosis or listeria infection,
* no previous history of cancer other than successfully treated skin cancer;
* women can not be pregnant or be breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000
Dates: Start 2002-09

PRIMARY OUTCOMES:
Change in disease activity score at visit week 12 as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: William M. Edwards, M.D., Principal Investigator — Low Country Research Center, North Charelston SC
Locations (54):
- United States (54):
  - Thomas McGee, MD, Mobile, Alabama
  - Desert Valley Medical, Apple Valley, California
  - Kenneth Hsu, MD, Inc., Bakersfield, California
  - Rheumatology Clinic, Los Angeles, California
  - Michael Harrington, MD, Napa, California
  - Midori Jane Nishio, MD, Walnut Creek, California
  - Naveen Raja, MD, Whittier, California
  - Mountain Rheumatology, Denver, Colorado
  - Division of Rheumatic Diseases/University of CT Health Center, Farmington, Connecticut
  - New Haven Medical Group, PC, New Haven, Connecticut
  - Norman Gaylis, MD, Aventura, Florida
  - Mike Schweitz, MD, West Palm Beach, Florida
  - Maurice McCarthy, MD, Winter Haven, Florida
  - Intermountain Orthopedics, Boise, Idaho
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Loyola University Medical Center, Maywood, Illinois
  - West Suburban Health Care, Oak Park, Illinois
  - OSF Medical Group -Rheumatology, Peoria, Illinois
  - Rockford Clinic, Clinical Research Department, Rockton, Illinois
  - Pain Therapy Center, Schaumburg, Illinois
  - Baton Rouge Clinic, Baton Rouge, Louisiana
  - Thomas Pressly, MD, Shreveport, Louisiana
  - Rheumatology Associates, Portland, Maine
  - Northampton Internal Medicine Association, Northampton, Massachusetts
  - Fallon Clinic Research, West Boylston, Massachusetts
  - John Howland, MD, Bay City, Michigan
  - Freeman Health Systems, Joplin, Missouri
  - Peggy Schlesinger, MD, Missoula, Montana
  - NJ Associates in Medicine, Fair Lawn, New Jersey
  - Internal Medicine and Rheumatic Diseases, Millburn, New Jersey
  - Placido Morano, MD, Brooklyn, New York
  - NYU Hospital for Joint Disease, New York, New York
  - Alan Kaell, MD, Port Jefferson Station, New York
  - Carolina Bone and Joint, PA, Monroe, North Carolina
  - Gordon Senter, MD Rheumatology, PA, Salisbury, North Carolina
  - MedCenter One Health Systems, Bismarck, North Dakota
  - University Hospital of Cleveland, Beachwood, Ohio
  - Arthritis Clinic, Canton, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - Arthritis and Osteoporosis Clinic, LLC, Bend, Oregon
  - Jel M. Depper, MD, Bend, Oregon
  - Sanford and Roumm Rheumatology, Camp Hill, Pennsylvania
  - Frederick Murphy, MD, Duncansville, Pennsylvania
  - Rheumatology Associates, Norristown, Pennsylvania
  - Rheumatology Associates, Ltd., Sellersville, Pennsylvania
  - Low Country Research Center, North Charleston, South Carolina
  - Medical Specialists of Nashville, Nashville, Tennessee
  - Arthritis and Osteoporosis Clinical Research Center of Central Texas, Waco, Texas
  - Center of Arthritis and Rheumatic Disease, PC, Chesapeake, Virginia
  - Margaret Gradzka, MD, Fairfax, Virginia
  - Metropolitan Clinical Research, Falls Church, Virginia
  - Northern Virginia Center for Arthritis, Reston, Virginia
  - Lewis-Gale Clinic, Salem, Virginia
  - ROAD Clinic, Lakewood, Washington

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778